CLINICAL TRIAL: NCT01857154
Title: A Double-Blinded Randomized Controlled CER Study of Changes in Bone Mineral Density, Blood Chemistries, Self-Reported Quality of Life and Compliance as a Function of Consuming Micronized Versus Non-micronized Calcium Carbonate
Brief Title: A Study of Changes in Bone Mineral Density as a Function of Consuming Two Different Forms of Calcium Carbonate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrative Health Technologies, Inc. (Network)
Responsible Party: Principal Investigator, Gilbert R Kaats, Dr. Gilbert R. Kaats, PhD, Integrative Health Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 064
Record Dates: First submitted 2013-05-08; First posted 2013-05-20 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Osteopenia, Osteoporosis
Keywords: Bone mineral density; Bone mineral content; Bone density; Bone health; Dual-energy x-ray absorptiometry
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bisphosphonates/Micronized Calcium Carbonate/Vitamin D3 (Active Comparator): Subjects currently being treated with Bisphosphonates will replace any calcium they are currently taking with four Capsules/Day containing a total amount of 500 mg of Micronized Calcium Carbonate and 800 IU Vitamin D3
  Interventions: Dietary Supplement: Micronized Calcium Carbonate; Dietary Supplement: Vitamin D3
- Bisphosphonates/Non-Micronized Calcium Carbonate/Vitamin D3 (Active Comparator): Subjects currently being treated with Bisphosphonates will replace any calcium they are currently taking with four Capsules/Day containing a total amount of 1000 mg of Non-Micronized Calcium Carbonate and 800 IU Vitamin D3.
  Interventions: Dietary Supplement: Non-Micronized Calcium Carbonate; Dietary Supplement: Vitamin D3
- Non-Micronized Calcium Carbonate/Vitamin D3 (Active Comparator): Subjects who are not currently being treated with Bisphosphonates will replace any calcium they are currently taking with four Capsules/Day containing a total of 1000 mg of Non-Micronized Calcium Carbonate and 800 IU Vitamin D3.
  Interventions: Dietary Supplement: Non-Micronized Calcium Carbonate; Dietary Supplement: Vitamin D3
- Micronized Calcium Carbonate/Vitamin D3 (Active Comparator): Subjects who are not currently being treated with Bisphosphonates will replace any calcium they are currently taking with four Capsules/Day containing a total of 500 mg of Micronized Calcium Carbonate and 800 IU Vitamin D3
  Interventions: Dietary Supplement: Micronized Calcium Carbonate; Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Micronized Calcium Carbonate — Subjects currently being treated with bisphosphonates will be administered 500 mg micronized calcium carbonate.
  Subjects not currently being treated with bisphosphonates will be administered 500 mg micronized calcium carbonate.
  Arms: Bisphosphonates/Micronized Calcium Carbonate/Vitamin D3; Micronized Calcium Carbonate/Vitamin D3
Dietary Supplement: Non-Micronized Calcium Carbonate — Subjects currently being treated with bisphosphonates will be administered 1000 mg non-micronized calcium carbonate.
  Subjects not currently being treated with bisphosphonates will be administered 1000 mg non- micronized calcium carbonate.
  Arms: Bisphosphonates/Non-Micronized Calcium Carbonate/Vitamin D3; Non-Micronized Calcium Carbonate/Vitamin D3
Dietary Supplement: Vitamin D3 — All subjects in the study cohort will be administered 800 IU Vitamin D3.

SUMMARY:
The purpose of this study is to determine whether consuming calcium carbonate that has been micronized is more effective than the traditional form of calcium carbonate in maintaining or increasing bone mineral density in people who are currently taking bisphosphonates or other bone-health medications.

DETAILED DESCRIPTION:
Addressing the need for a form of supplemental calcium that could facilitate increases in BMD without the adverse effects often reported with limestone-based forms of calcium, a patented technology was developed to increase calcium absorbability using both Zet Mill/Ball Mill bottom-up pulverizing technology and 4D top-down ebonite charging technology to create a novel form of calcium referred to as micronized calcium carbonate (MCC). In comparison to other technologies that use water and high heat, which results in a loss of core nutrients and decreased product efficacy, the calcium produced by this unique pulverizing technology is micron-sized (0.03um - 10um) and therefore believed to be more effective. While its tiny size was thought to increase its absorption, the belief was that the intense activation of zinc via the patented ebonite charging process that could maximize the bioavailability of this calcium.

ELIGIBILITY:
Inclusion Criteria:

* Must currently be under the care of a physician and taking prescription medication for bone health
* Must ensure with medical provider that there are no medical conditions that would preclude participation
* Must be able to swallow capsules
* Must be age 21 or above
* Must agree to follow study requirements as set forth in Informed Consent

Exclusion Criteria:

* Men and women not currently taking prescription medication for bone health
* Conditions that inhibit gastrointestinal absorption of supplements
* Men and women less than 21 years of age
* Pregnant or breast feeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Bone Mineral Density as a measurement by Dual Energy X-ray Absorptiometry | 0 and 183 days
  Bone density scanning, also called dual-energy x-ray absorptiometry (DXA) or bone densitometry, is an enhanced form of x-ray technology that is used to measure bone mineral density. Imaging with x-rays involves exposing a part of the body to a small dose of ionizing radiation to produce pictures of the inside of the body.
  Benefits
  * DXA bone densitometry is a simple, quick and noninvasive procedure.
  * No anesthesia is required.
  * The amount of radiation used is extremely small-less than one-tenth the dose of a standard chest x-ray, and less than a day's exposure to natural radiation.
  * DXA bone density testing is the most accurate method available for the diagnosis of osteoporosis and is also considered an accurate estimate

SECONDARY OUTCOMES:
Blood Chemistry Panel | 0 and 183 days
  43 chemistries including lipids, Complete Blood Count, metabolic panel, Thyroid Stimulating Hormone and Cardio C-reactive Protein
Systolic and Diastolic blood pressure | 0 and 183 days
  Measures the amount of force (pressure) that blood exerts on the walls of blood vessels as it passes through them. Systolic blood pressure is a measure of blood pressure while the heart is beating. Diastolic pressure is a measure of blood pressure while the heart is relaxed, between heartbeats. Measurements will be taken after lying down for at least 5 minutes. Changes will be reported between baseline and day 183 of study.
Resting heart rate | 0 and 183 days
  Measure of heart rate after lying down for at least 5 minutes. Changes will be reported between baseline and day 183 of study.
Self-reported quality of life | 0 and 183 days
Number of participants with adverse effects | up to 183 days
  Participants will have opportunity to report on a weekly basis an adverse effects experienced

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert R Kaats, PhD FACN, Principal Investigator — Integrative Health Technologies, Inc.; Harry G Preuss, MD MACN, Study Chair — Georgetown University Medical Center, Dept of Biochemistry, Medicine and Pathology; Sidney J Stohs, PhD, Study Director — Dean Emeritus, Creighton University Health Sciences Center
Locations (1):
- Integrative Health Technologies, San Antonio, Texas, United States